CLINICAL TRIAL: NCT03503851
Title: Noninferiority Trial of MitraClip Implantation Strategies: 1 Clip vs. 2 Clips in Patients With Functional Mitral Regurgitation (One-Plus-One)
Brief Title: Noninferiority Trial of MitraClip Implantation Strategies: 1 Clip vs. 2 Clips in Patients With Functional Mitral Regurgitation
Acronym: One-Plus-One
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Delay during study initiation. Change of MitraClip design in meantime.
Sponsor: Asklepios proresearch (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #3150
Record Dates: First submitted 2018-03-06; First posted 2018-04-20 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Mitral Regurgitation Functional
Keywords: Mitral Regurgitation; transcatheter mitral valve repair; MitraClip
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, randomized, parallel-arm trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One CLIP (Active Comparator): Implantation of single MitraClip
  Interventions: Device: MitraClip implantation
- Two CLIPs (Active Comparator): Implantation of second MitraClip (after successful Implantation of single MitraClip)
  Interventions: Device: MitraClip implantation

INTERVENTIONS:
Device: MitraClip implantation — Device to approximate the mitral valve leaflets

SUMMARY:
Implantation of the MitraClip has become the most frequently used percutaneous technique to treat significant (grade 3+ or 4+) mitral regurgitation (MR) in elderly patients deemed inoperable or at high surgical risk. In Europe, about two-thirds of patients treated with the MitraClip suffer from MR of functional origin secondary to ischemic or dilated cardiomyopathy. At present, there is debate among operators on whether stabilizing/supporting a single adequately implanted clip with a second clip is beneficial for patients with functional MR.

DETAILED DESCRIPTION:
Implantation of the MitraClip has become the most frequently used percutaneous technique to treat significant (grade 3+ or 4+) mitral regurgitation (MR) in elderly patients deemed inoperable or at high surgical risk. In Europe, about two-thirds of patients treated with the MitraClip suffer from MR of functional origin secondary to ischemic or dilated cardiomyopathy. At present, there is debate among operators on whether stabilizing/supporting a single adequately implanted clip with a second clip is beneficial for patients with functional MR.

Purpose To demonstrate the noninferiority of a 1-clip strategy vs. a 2-clip strategy of MitraClip implantation, when the second clip in the 2-clip study arm is implanted for stabilizing/supporting purposes.

ELIGIBILITY:
Inclusion Criteria:

* Absence of a structural abnormality of the mitral valve giving rise to MR.
* MR severity of US grade 3+ or 4+ of central or noncentral origin
* Patient must consent to randomization in the hybrid operating theater upon successful implantation of a single MitraClip. Written informed consent must be provided prior to the MitraClip procedure.

Exclusion Criteria:

* patients with primary regurgitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of number of participants who died death within one year | 1 year
  death
Evaluation of number of rehospitalizations due to heart failure among patients receiving one or two clips | 1 year
  heart failure rehospitalization
Evaluation of number of participants with recurrent regurgitation within one year | 1 year
  recurrence of mitral regurgitation (>grade 2+ at 1 year)

SECONDARY OUTCOMES:
death | 1 year
  freedom from death (1-year)
heart failure | 1 year
  freedom from heart failure (1-year)
rehospitalization | 1-year
  rehospitalization
regurgitation | 1-year
  freedom from recurrence of mitral regurgitation (>2+; 1-year)
success rate | 1-year
  procedural success rate in 2-clip arm
procedure duration | 1-year
  procedure duration
total device time | 1-year
  total device time
fluoroscopy time | 1-year
  fluoroscopy time
contrast volume | 1-year
  contrast volume
complications | 1-year
  periprocedural (30-day) complications
echocardiographic variables | 1-year
  The following echocardiographic variables will be assessed by 2-dimensional transthoracic echocardiography at 12 months: Left ventricular (LV) end-diastolic diameter and volume; LV end-systolic diameter and volume; LV ejection fraction; LV outflow tract diameter and velocity time integral in LV outflow tract (to calculate forward stroke volume).
changes in echocardiographic variables | 1-year
  Changes from baseline to 12 months in echocardiographically assessed (at both time points) LV end-diastolic diameter and volume; LV end-systolic diameter and volume; LV ejection fraction; and forward stroke volume.
NYHA | 1-year
  NYHA functional class
6-minutes walk | 1-year
  6-minutes walk distance
quality of life | 1-year
  Assessment of the Minnesota Living With Heart Failure Questionnaire (MLHFQ) quality-of-life score. The questionnaire consists of 21 quality-of-life questions to be answered by the patient on a grading scale of 0 (best) to 5 (worst). Thus, the overall MLHFQ score ranges from 0 to 105.

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, MD, PHD, Principal Investigator — Asklepios Klinik St. Georg, Dept. of Cardiology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feldman T, Kar S, Elmariah S, Smart SC, Trento A, Siegel RJ, Apruzzese P, Fail P, Rinaldi MJ, Smalling RW, Hermiller JB, Heimansohn D, Gray WA, Grayburn PA, Mack MJ, Lim DS, Ailawadi G, Herrmann HC, Acker MA, Silvestry FE, Foster E, Wang A, Glower DD, Mauri L; EVEREST II Investigators. Randomized Comparison of Percutaneous Repair and Surgery for Mitral Regurgitation: 5-Year Results of EVEREST II. J Am Coll Cardiol. 2015 Dec 29;66(25):2844-2854. doi: 10.1016/j.jacc.2015.10.018. PMID 26718672
- [Background] Feldman T, Foster E, Glower DD, Kar S, Rinaldi MJ, Fail PS, Smalling RW, Siegel R, Rose GA, Engeron E, Loghin C, Trento A, Skipper ER, Fudge T, Letsou GV, Massaro JM, Mauri L; EVEREST II Investigators. Percutaneous repair or surgery for mitral regurgitation. N Engl J Med. 2011 Apr 14;364(15):1395-406. doi: 10.1056/NEJMoa1009355. Epub 2011 Apr 4. PMID 21463154
- [Background] Franzen O, Baldus S, Rudolph V, Meyer S, Knap M, Koschyk D, Treede H, Barmeyer A, Schofer J, Costard-Jackle A, Schluter M, Reichenspurner H, Meinertz T. Acute outcomes of MitraClip therapy for mitral regurgitation in high-surgical-risk patients: emphasis on adverse valve morphology and severe left ventricular dysfunction. Eur Heart J. 2010 Jun;31(11):1373-81. doi: 10.1093/eurheartj/ehq050. Epub 2010 Mar 10. PMID 20219746
- [Background] Baldus S, Schillinger W, Franzen O, Bekeredjian R, Sievert H, Schofer J, Kuck KH, Konorza T, Mollmann H, Hehrlein C, Ouarrak T, Senges J, Meinertz T; German Transcatheter Mitral Valve Interventions (TRAMI) investigators. MitraClip therapy in daily clinical practice: initial results from the German transcatheter mitral valve interventions (TRAMI) registry. Eur J Heart Fail. 2012 Sep;14(9):1050-5. doi: 10.1093/eurjhf/hfs079. Epub 2012 Jun 8. PMID 22685268
- [Background] Grasso C, Capodanno D, Scandura S, Cannata S, Imme S, Mangiafico S, Pistritto A, Ministeri M, Barbanti M, Caggegi A, Chiaranda M, Dipasqua F, Giaquinta S, Occhipinti M, Ussia G, Tamburino C. One- and twelve-month safety and efficacy outcomes of patients undergoing edge-to-edge percutaneous mitral valve repair (from the GRASP Registry). Am J Cardiol. 2013 May 15;111(10):1482-7. doi: 10.1016/j.amjcard.2013.01.300. Epub 2013 Feb 20. PMID 23433761
- [Background] Surder D, Pedrazzini G, Gaemperli O, Biaggi P, Felix C, Rufibach K, der Maur CA, Jeger R, Buser P, Kaufmann BA, Moccetti M, Hurlimann D, Buhler I, Bettex D, Scherman J, Pasotti E, Faletra FF, Zuber M, Moccetti T, Luscher TF, Erne P, Grunenfelder J, Corti R. Predictors for efficacy of percutaneous mitral valve repair using the MitraClip system: the results of the MitraSwiss registry. Heart. 2013 Jul;99(14):1034-40. doi: 10.1136/heartjnl-2012-303105. Epub 2013 Jan 23. PMID 23343688
- [Background] Maisano F, Franzen O, Baldus S, Schafer U, Hausleiter J, Butter C, Ussia GP, Sievert H, Richardt G, Widder JD, Moccetti T, Schillinger W. Percutaneous mitral valve interventions in the real world: early and 1-year results from the ACCESS-EU, a prospective, multicenter, nonrandomized post-approval study of the MitraClip therapy in Europe. J Am Coll Cardiol. 2013 Sep 17;62(12):1052-1061. doi: 10.1016/j.jacc.2013.02.094. Epub 2013 Jun 7. PMID 23747789
- [Background] Nickenig G, Estevez-Loureiro R, Franzen O, Tamburino C, Vanderheyden M, Luscher TF, Moat N, Price S, Dall'Ara G, Winter R, Corti R, Grasso C, Snow TM, Jeger R, Blankenberg S, Settergren M, Tiroch K, Balzer J, Petronio AS, Buttner HJ, Ettori F, Sievert H, Fiorino MG, Claeys M, Ussia GP, Baumgartner H, Scandura S, Alamgir F, Keshavarzi F, Colombo A, Maisano F, Ebelt H, Aruta P, Lubos E, Plicht B, Schueler R, Pighi M, Di Mario C; Transcatheter Valve Treatment Sentinel Registry Investigators of the EURObservational Research Programme of the European Society of Cardiology. Percutaneous mitral valve edge-to-edge repair: in-hospital results and 1-year follow-up of 628 patients of the 2011-2012 Pilot European Sentinel Registry. J Am Coll Cardiol. 2014 Sep 2;64(9):875-84. doi: 10.1016/j.jacc.2014.06.1166. PMID 25169171
- [Background] Eggebrecht H, Schelle S, Puls M, Plicht B, von Bardeleben RS, Butter C, May AE, Lubos E, Boekstegers P, Ouarrak T, Senges J, Schmermund A. Risk and outcomes of complications during and after MitraClip implantation: Experience in 828 patients from the German TRAnscatheter mitral valve interventions (TRAMI) registry. Catheter Cardiovasc Interv. 2015 Oct;86(4):728-35. doi: 10.1002/ccd.25838. Epub 2015 Feb 12. PMID 25601532
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed